CLINICAL TRIAL: NCT02814019
Title: A Phase III Double-blind, Randomized, Placebo-Controlled Study Assessing the Efficacy, Safety and Tolerability of Idebenone in Patients With Duchenne Muscular Dystrophy Receiving Glucocorticoid Steroids
Brief Title: A Phase III Double-blind Study With Idebenone in Patients With Duchenne Muscular Dystrophy (DMD) Taking Glucocorticoid Steroids
Acronym: SIDEROS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis concluded to futility
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-III-012
Record Dates: First submitted 2016-06-17; First posted 2016-06-27 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: respiratory function in DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- idebenone 150 mg film-coated tablets (Experimental): 900 mg idebenone/day (2 tablets to be taken 3 times a day with meals)
  Interventions: Drug: Idebenone 150 mg film-coated tablets
- placebo (Placebo Comparator): matching placebo tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Idebenone 150 mg film-coated tablets
  Arms: idebenone 150 mg film-coated tablets
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to assess the efficacy of idebenone in delaying the loss of respiratory function in patients with DMD receiving concomitant glucocorticoid steroids

DETAILED DESCRIPTION:
The SIDEROS trial is a randomized, placebo controlled, parallel group study of the efficacy of idebenone in delaying the loss of respiratory function, whilst also monitoring safety and tolerability of idebenone in at least 266 DMD patients taking stable dose of concomitant glucocorticoid steroids.

The study treatment period will be 18 months/ 78 weeks and the idebenone dose will be 900 mg/day. Participants can use deflazacort or prednisolone and be on any dose regimen.

Since glucocorticoid steroids are widely used in ambulant boys from an early age until late into teenage and even adult years, this study will not take age and ambulatory status into account and will only exclude patients that need daytime ventilator assistance.

The schedule of assessments will include a Screening Visit and up to 9 protocol visits, including a Follow-up Visit.

A Screening Visit will take place a maximum of 4 weeks prior to the Baseline Visit (Visit 1, study day -1). Beginning at Baseline, the patient will receive study medication to be taken at home, and will undergo regular assessments in the clinic throughout the study period until Visit 8 at Week 78 at which time the study will be completed and medication discontinued.

All patients completing Visit 8/Week 78, and considered eligible by the Investigator will be able to participate in an open-label extension study (SIDEROS-E) and will continue to receive idebenone until idebenone is commercially available for patients included in the study or SIDEROS-E is terminated by the Sponsor, whichever occurs first. The duration of the SIDEROS-E study will be defined in a separate protocol.

For all patients not participating in the extension study (SIDEROS-E), a Follow-up Visit (Visit 9/Follow-up Visit) will take place 4 weeks after end of Treatment at Visit 8/Week 78 or after premature discontinuation of study medication.

Each hospital visit will include efficacy assessments (respiratory function assessed by hospital-based spirometry, oxygen saturation, end-tidal CO2) and safety assessments (adverse events, concomitant medication, physical examination, vital signs, safety laboratory evaluations). In addition, respiratory function will be assessed weekly at home with a hand-held device in order to closely monitor respiratory function between hospital visits.

The study medication, all medical procedures and laboratory testing, and the visits to the study centre are free of charge. In addition the patients will receive a travel allowance to cover reasonable expenses to and from the study centre. Participants will not otherwise be compensated for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with a 35% ≤ FVC ≤ 80% of predicted value at Screening and at Baseline and who, in the opinion of the investigator are in the respiratory function decline phase.
2. Minimum 10 years old at Screening.
3. Signed and dated Informed Consent Form.
4. Documented diagnosis of DMD (severe dystrophinopathy) and clinical features consistent of typical DMD at diagnosis (i.e. documented delayed motor skills and muscle weakness by age 5 years). DMD should be confirmed by mutation analysis in the dystrophin gene or by substantially reduced levels of dystrophin protein (i.e. absent or <5% of normal) on Western blot or immunostaining.
5. Chronic use of systemic glucocorticoid steroids for DMD related conditions continuously for at least 12 months prior to Baseline without any dose adjustments on a mg/kg basis in the last 6 months (only dose adjustments determined by weight changes are allowed).
6. Ability to provide reliable FVC values at Screening and Baseline, and reproducible within 15% (relative change) at Baseline compared to Screening.
7. Patients assessed by the Investigator as willing and able to comply with the requirements of the study, possess the required cognitive abilities and are able to swallow study medication.
8. Patients who prior to Screening have been immunized with 23-valent pneumococcal polysaccharide vaccine or any other pneumococcal polysaccharide vaccine as per national recommendations, as well as annually immunized with inactivated influenza vaccine.

Exclusion Criteria:

1. Symptomatic heart failure (defined as patients with structural heart disease, dyspnea, fatigue and impaired tolerance to exercise; Stage C by the ACCF/AHA guideline or NYHA Classes III-IV) and/or symptomatic ventricular arrhythmias.
2. Ongoing participation in any other therapeutic trial and/or intake of any investigational drug within 90 days prior to Baseline (only exception allowed is use of Deflazacort in the US as part of the Expanded Access Program, or any approved corticosteroid product in trial for regimen optimization, for which the patient met the inclusion criterion 5).
3. Ongoing exon-skipping therapy or read-through gene therapy for DMD; previous exon-skipping or read-through gene therapy is allowed if the stop date was more than 6 months prior to Screening.
4. Planned or expected spinal fusion surgery during the study period (as judged by the Investigator; i.e. due to rapidly progressing scoliosis), previous spinal fusion surgery is allowed if it took place more than 6 months prior to Screening.
5. Asthma, bronchitis/COPD, bronchiectasis, emphysema, pneumonia or presence of any other non-DMD respiratory illness that affects respiratory function.
6. Chronic use of beta2-agonists or any use of other bronchodilating/bronchoconstricting medication (inhaled steroids, sympathomimetics, anticholinergics, antihistamines); chronic use is defined as a daily intake for more than 14 days.
7. Any bronchopulmonary illness that required treatment with antibiotics within 3 months prior to Screening.
8. Moderate or severe hepatic impairment (use as guidance Child-Pugh class B [7 to 9 points] or Child-Pugh class C [10 to 15 points] - see Appendix B) or severe renal impairment (eGFR <30 mL/min/1.73 m2).
9. Prior or ongoing medical condition or laboratory abnormality that in the Investigator's opinion may put the patient at significant risk may confound the study results or may interfere significantly with the patient's participation in the study.
10. Relevant history of or current drug or alcohol abuse, or use of any tobacco or marijuana products/smoking.
11. Known individual hypersensitivity to idebenone or to any of the ingredients or excipients of the study medication.
12. Daytime ventilator assistance (defined as use of any assisted ventilation while awake).

Note: Patients who suffer from a severe, unstable condition including (but not limited to) cancer, auto-immune diseases, hematological diseases, metabolic disorders or immunodeficiencies, and who are at risk of an aggravation unrelated to the study condition, can only be included in the study if accepted in writing by the Sponsor's Senior Clinical Research Physician.

Min Age: 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Forced Vital Capacity percent predicted (FVC %p) at Week 78 | 78 weeks
  Delaying the loss of respiratory function in patients with DMD receiving glucocorticoid steroids as measured by changes in FVC %p from Baseline to Week 78 using hospital based spirometry.

SECONDARY OUTCOMES:
Change From Baseline in Percent Predicted Peak Expiratory Flow (PEF %p) at Week 78 | 78 weeks
  Delaying the loss of respiratory function in patients with DMD receiving glucocorticoid steroids as measured by:
  •The change from Baseline to Week 78 in PEF %p assessed by hospital-based spirometry measurements
Change From Baseline in Forced Vital Capacity (FVC) at Week 78 | 78 weeks
  Delaying the loss of respiratory function in patients with DMD receiving glucocorticoid steroids as measured by:
  •The time to first 10% decline in FVC (L) during the 78-week treatment period, assessed by hospital-based spirometry measurements
Change from Baseline in Inspiratory Flow Reserve (IFR) at Week 78 | 78 weeks
  Delaying the loss of respiratory function in patients with DMD receiving glucocorticoid steroids as measured by:
  •The change from Baseline to Week 78 in IFR assessed by hospital-based spirometry measurements

CONTACTS AND LOCATIONS:
Locations (63):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Department of Physical Medicine and Rehabilitation, Sacramento, California
  - Loma Linda University Healthcare, San Bernardino, California
  - Shriners Hospitals for Children-Tampa, Tampa, Florida
  - Rare Disease Research, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Fairway, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Neurosciences Institute, Neurology - Charlotte Carolinas Healthcare System, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Gottfried von Preyer'sches Kinderspital, Vienna, Austria
- Belgium (2):
  - University Hospital Leuven, Leuven
  - Centre de Référence Neuromusculaire, CHR Citadelle, Liège
- Sofia Medical University, Sofia, Bulgaria
- France (5):
  - Service de neuropédiatrie Pôle Pédiatrie CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Hôtel Dieu, Nantes
  - I-Motion - Plateforme d'essais cliniques pédiatriques Hôpital Armand Trousseau bâtiment Lemariey porte 20, Paris
  - Hôpital des enfants, Toulouse
- Germany (7):
  - Universitätsmedizin Berlin Campus Virchow-Klinikum, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Universitätsklinik Freiburg Zentrum für Kinderheilkunde und Jugendmedizin, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Kinder- und Jugendmedizin, Hamburg
  - Universitätsklinikum Heidelberg Zentrum für Kinder- und Jugendmedizin, Heidelberg
  - Zentrum für neuromuskuläre Erkrankungen, München
- Semmelweis University 2nd Department of Paediatrics, Budapest, Hungary
- Children's University Hospital, Dublin, Ireland
- Institute of Neurology at Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Italy (8):
  - Fondazione IRCCS Eugenio Medea, Bosisio Parini
  - Istituto Giannina Gaslini, Genova
  - Scientific Coordinator Nemo Sud Clinical Center, Messina
  - Centro Clinico NEMO (NEuroMuscular Omnicentre), Niguarda Hospital, Milan
  - Servizio di Cardiomiologia e Genetica Medica, AOU Università degli Studi della Campania "Luigi Vanvitelli", Napoli
  - Reparto Di Neurologia dell'Osperdale Di Padova, Padua
  - Dipartimento di Clinica Neurologica e Psichiatrica dell'Età Evolutiva della Fondazione IRCCS "C. Mondino" di Pavia, Pavia
  - U.O.C. Neuropsichiatria Infantile, Roma
- Netherlands (2):
  - LUMC, Leiden
  - Radboud university medical centre, Nijmegen
- Spain (5):
  - Hospital Sant Joan de Déu Neuropediatra, Barcelona
  - Hospital Universitari Vall D' Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital La Fe de Valencia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Center for neuromuscular disorders, Universitäts-Kinderspital beider Basel (UKBB), Basel, Switzerland
- United Kingdom (7):
  - Leeds Teaching Hospital NHS Trust, Leeds
  - UCL, National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital for Children, London
  - John Walton Muscular Dystrophy Research Centre, Newcastle
  - Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry
  - Oxford University hospitals NHS Foundation Trust, Oxford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] Buyse GM, Voit T, Schara U, Straathof CSM, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, McDonald CM, Rummey C, Meier T; DELOS Study Group. Efficacy of idebenone on respiratory function in patients with Duchenne muscular dystrophy not using glucocorticoids (DELOS): a double-blind randomised placebo-controlled phase 3 trial. Lancet. 2015 May 2;385(9979):1748-1757. doi: 10.1016/S0140-6736(15)60025-3. Epub 2015 Apr 20. PMID 25907158
- [Background] McDonald CM, Meier T, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Spagnolo P, Buyse GM; DELOS Study Group. Idebenone reduces respiratory complications in patients with Duchenne muscular dystrophy. Neuromuscul Disord. 2016 Aug;26(8):473-80. doi: 10.1016/j.nmd.2016.05.008. Epub 2016 May 12. PMID 27238057
- [Background] Buyse GM, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Mayer OH, Spagnolo P, Meier T, McDonald CM; DELOS Study Group. Treatment effect of idebenone on inspiratory function in patients with Duchenne muscular dystrophy. Pediatr Pulmonol. 2017 Apr;52(4):508-515. doi: 10.1002/ppul.23547. Epub 2016 Aug 29. PMID 27571420